CLINICAL TRIAL: NCT06921005
Title: Can Lower-body Occlusion During Low-intersity Cycling Influence Recovery of Youth Elite Soccer Players?
Brief Title: Can Lower-body Occlusion Influence Sports Recovery?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Filipe Silvano Pinto Maia, Principal Investigator, University of Maia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: ST_PhD_01
Record Dates: First submitted 2025-02-24; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Recovery of Function; Sports
Keywords: sports; recovery; blood flow restriction
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- AR (Experimental): Active recovery group
  Interventions: Other: Exercise
- AR+ continuous BFR (Experimental): Active recovery group with continuous blood flow restriction
  Interventions: Other: Exercise
- AR + intermittent BFR (Experimental): Actve recovery group with intermittent blood flow restriction
  Interventions: Other: Exercise
- Control group (Active Comparator): Control group
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Recovery with vascular occlusion or active recovery in soccer players.

SUMMARY:
This study ai ms to compare the recovery kinetics of different interventions: i) active recovery; ii) continuous vascular occlusion during active recovery; iii) intermittent vascular occlusion during active recovery; iv) control group.

ELIGIBILITY:
Inclusion Criteria:

* soccer players
* elite athletes
* present in the pitch training sessions

Exclusion Criteria:

* injured athletes
* female athletes

Ages: 17 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
countermovement jump height | Baseline, post 30 minutes, post 24 hours
  countermovement jump height measured using chronojump.
squat jump height | Baseline, post 30 minutes, post 24 hours
  Squat jump height measured using chronojump
Bar velocity during squat | Baseline, post 30 minutes, post 24 hours
  Squat velocity measured using a linear encoder
hip thrust bar velocity | Baseline, post 30 minutes, post 24 hours
  hip thrust bar velocity measured using a linear encoder
Perceived fatigue | Baseline, post 30 minutes, and post 24 hours.
  Perceived fatigue measured using the Rating of Fatigue Scale (range: 0 - 10)
Muscle soreness Visual Analogue Scale | Baseline, 30 minutes post, 24 hours post.
  Muscle soreness measured using a Visual Analogue Scale (0 - 10)
Perceived recovery | Baseline, 30 minutes post, 24 hours post.
  Perceived recovery measured using the Total Quality Recovery Scale (range 6 - 20)

IPD SHARING:
Plan to Share IPD: Undecided